CLINICAL TRIAL: NCT03345550
Title: Pilot Study of Omega-3 Polyunsaturated Fatty Acid Treatment in Mild Acute TBI (OPTIMA-TBI Pilot)
Brief Title: OPTIMA-TBI Pilot Study
Acronym: OPTIMA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual of patients, lack of financial resources
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Frederick Korley, MD, PhD, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00129045
Record Dates: First submitted 2017-11-12; First posted 2017-11-17 (Actual); Results first posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-04

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion | interventions — Docosahexaenoic Acids; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Omega-3 Polyunsaturated Fatty Acid Treatment Arm (Experimental): Participants randomized to this study arm will receive 6g DHA+EPA for one month followed by 1.2 g DHA+EPA for two months. Capsules contain fish oil 1000 mg (contains 500 mg DHA & 100 mg EPA) or placebo capsules.
  Interventions: Drug: Omega-3 Polyunsaturated Fatty Acids (Fish Oil 1000 mg (contains 500 mg DHA & 100 mg EPA)) or placebo capsules.
- Placebo Arm (Placebo Comparator): Participants randomized to this study arm will receive placebo drug for 3 months.
  Interventions: Drug: Placebo - Cap

INTERVENTIONS:
Drug: Omega-3 Polyunsaturated Fatty Acids (Fish Oil 1000 mg (contains 500 mg DHA & 100 mg EPA)) or placebo capsules. — Participants will be randomized to receive fish oil 1000 mg (contains 500 mg DHA & 100 mg EPA) or placebo capsules.
  Arms: Omega-3 Polyunsaturated Fatty Acid Treatment Arm
Drug: Placebo - Cap — Participants will be randomized to receive fish oil 1000 mg (contains 500 mg DHA & 100 mg EPA) or placebo capsules (olive oil capsules that look identical to the intervention DHA+EPA).
  Arms: Placebo Arm

SUMMARY:
This is a double-blind, randomized controlled trial comparing the effect of omega-3 fatty acid versus placebo on blood biomarkers of brain injury, inflammation and neurogenesis.

DETAILED DESCRIPTION:
Primary brain injury, the initial physical injury to brain tissue post-trauma, responds only to measures that prevent TBI from occurring in the first place. However, secondary brain injury, a complex cascade of events causing additional brain injury following primary brain injury, is more amenable to pharmacologic treatment. Neuroinflammation is one of the recognized mechanisms of secondary brain injury. In response to primary brain injury, activated microglia and injured neurons both release signaling proteins including cytokines and chemokines. Ω-3 and ω-6 fatty acids are major components of immune cells and neuronal cell membranes. They are also precursors to neuromodulatory lipids such as eicodanoids, endovanilloids and endocannabinoids that have antinociceptive and anxiolytic properties. Docosahexaenoic acid (DHA) is one of the most abundant fatty acid components of brain cell membrane phospholipids. In rodent model studies, dietary supplementation with omega-3 fatty acids (eicosapentaenoic acid [EPA] and docosahexaenoic acid [DHA]) decreased secondary axonal injury, attenuated endoplasmic reticulum stress response, decreased neuroinflammation post-TBI, and improved short and long-term neurologic outcomes. Additionally, DHA supplementation post-TBI enhances neurogenesis by counteracting reductions in neuroplasticity biomarkers such as brain-derived neurotrophic factor. Furthermore, DHA deficient rodents are more likely to have a greater amount of axonal injury and slower recovery neurologic recovery post-TBI. To our knowledge there are no human studies examining the effect of omega-3 fatty acid supplementation post-TBI on functional, symptomatic and neurologic outcomes. However, a study of collegiate football players who were randomized to 2, 4 or 6g/day of DHA or placebo for a total of 189 days (including 80 pre-season days). Irrespective of the dose of DHA supplementation, those receiving DHA had lower values of serum neurofilament light chain, a biomarker of axonal injury, than those receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Individuals presenting to the emergency department (ED) within 24 hours of injury, who meet the American Congress of Rehabilitation Medicine (ACRM)'s definition of having mild traumatic brain injury (mTBI) will be eligible
* The ACRM defines mTBI as a traumatically-induced physiological disruption of brain function as a consequence of the head being struck, striking an object, or undergoing an acceleration/deceleration movement without direct external head trauma and resulting in at least one of the following:
* any period of loss of consciousness (LOC)
* any loss of memory for events immediately before or after the injury
* any alteration in mental state at the time of the injury (eg, feeling dazed, disoriented, or confused)
* focal neurological deficit(s) that may or may not be transient

Exclusion Criteria:

* GCS<13 at any time during ED stay.
* Significant polytrauma including: bony fracture or solid organ injury
* Study medication cannot be administered within 24 hours of injury
* Patient cannot be relied on to complete follow-up (i.e. no reliable telephone number, substance dependence, homeless)
* Cannot communicate in English
* Take an anticoagulant (coumadin or a novel oral anticoagulant) daily
* Age less than 18 years or greater than 65 years
* Patients already taking fish oil supplements daily
* History of cognitive impairment
* Allergic to fish/fish oil
* Pregnant women (self-reported)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Korley, M.D., Ph.D., Principal Investigator — Department of Emergency Medicine
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Omega-3 Polyunsaturated Fatty Acid Treatment Arm: Participants randomized to this study arm received 6g DHA+EPA for one month followed by 1.2 g DHA+EPA for two months. Capsules contain fish oil 1000 mg (contains 500 mg DHA & 100 mg EPA) or placebo capsules.
  Omega-3 Polyunsaturated Fatty Acids (Fish Oil 1000 mg (contains 500 mg DHA & 100 mg EPA)) or placebo capsules.: Participants were randomized to receive fish oil 1000 mg (contains 500 mg DHA & 100 mg EPA) or placebo capsules.
- Placebo Arm: Participants randomized to this study arm received placebo drug for 3 months.
  Placebo - Cap: Participants were randomized to receive fish oil 1000 mg (contains 500 mg DHA & 100 mg EPA) or placebo capsules (olive oil capsules that look identical to the intervention DHA+EPA).
Period: Overall Study
Arm/Group | Omega-3 Polyunsaturated Fatty Acid Treatment Arm | Placebo Arm
Started | 22 | 22
First Received Drug | 22 | 22
Completed | 17 | 17
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 Polyunsaturated Fatty Acid Treatment Arm | Placebo Arm | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37.5 [24.8 to 46.5] | 26.5 [22.8 to 38.5] | 30.5 [23.2 to 43.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 20 | 21 | 41
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 1 | 4 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 19 | 14 | 33
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Biomarker Endpoints (NFL)
Description: Neuronal injury measured by Neurofilament Light Chain (NFL). Samples will be analyzed using a digital immunoassay based on a single molecule counting technology.
Time Frame: Baseline,3 months
Population: For some of the assays, some individuals' data was not available.
Measure: Median (Inter-Quartile Range); unit: picograms per ml
Arm/Group | Omega-3 Polyunsaturated Fatty Acid Treatment Arm | Placebo Arm
Number analyzed (Participants) | 19 | 19
picograms per ml
  NFL baseline | 7.9 [5.1 to 11.4] | 5.3 [4.4 to 10.0]
  NFL 1 month: number analyzed (Participants) | 14 | 10
  NFL 1 month | 6.7 [3.9 to 12.7] | 8.7 [4.8 to 13.4]
  NFL 3 months: number analyzed (Participants) | 12 | 8
  NFL 3 months | 8.2 [4.1 to 9.5] | 9.7 [4.6 to 20.0]
Statistical Analysis 1: Comparison: Omega-3 Polyunsaturated Fatty Acid Treatment Arm vs Placebo Arm; Baseline; Test type: Superiority; p = .24, Kruskal-Wallis
Statistical Analysis 2: Comparison: Omega-3 Polyunsaturated Fatty Acid Treatment Arm vs Placebo Arm; 1 month analysis; Test type: Superiority; p = .43, Kruskal-Wallis
Statistical Analysis 3: Comparison: Omega-3 Polyunsaturated Fatty Acid Treatment Arm vs Placebo Arm; 3 month; Test type: Superiority; p = .54, Kruskal-Wallis

2. Primary Outcome: Biomarker Endpoint (Inflammation)
Description: We will measure serum levels of high sensitivity C-Reactive Protein (CRP)
Time Frame: 3 months
Population: While serum was collected no CRP data or measurements were made or can be made now or in the future.
Arm/Group | Omega-3 Polyunsaturated Fatty Acid Treatment Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Biomarker Endpoint (Neurogenesis)
Description: Serum levels of brain derived neurotrophic factor (BDNF)
Time Frame: 3 months
Population: While serum was collected, no BDNF data or measurements were collected or can be made now or in the future.
Arm/Group | Omega-3 Polyunsaturated Fatty Acid Treatment Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Delayed Functional Recovery
Description: Delayed functional recovery will be defined as a Glasgow Outcome Scale Extended (GOSE) <8 at 3 months. Scores range from 1-8. 8 is Upper good recovery and 1 is death
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Omega-3 Polyunsaturated Fatty Acid Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 17
Participants
  Upper good recovery at 3 months (GOSE=8) | 16 | 17
  Lower good recovery at 3 months (GOSE=7) | 1 | 0
Statistical Analysis 1: Comparison: Omega-3 Polyunsaturated Fatty Acid Treatment Arm vs Placebo Arm; Test type: Superiority; p = .31, Chi-squared

5. Secondary Outcome: Gastrointestinal Distress
Description: GI distress is measured by number of individuals who experienced it.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Omega-3 Polyunsaturated Fatty Acid Treatment Arm | Placebo Arm
Number analyzed (Participants) | 22 | 22
Participants | 3 | 0

6. Secondary Outcome: Clinically Significant Bleeding
Description: Clinically significant bleeding distress is measured by number of individuals who experienced it.
Time Frame: 3 months
Population: All 22 participants were analyzed on an Intention to Treat analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Omega-3 Polyunsaturated Fatty Acid Treatment Arm | Placebo Arm
Number analyzed (Participants) | 22 | 22
Participants | 0 | 0

7. Other Pre Specified Outcome: Cognitive Impairment
Description: Cognitive impairment will be defined by a battery of neurocognitive tests including the Montreal Cognitive Assessment (MOCA), Hopkins Verbal Learning Test (HVLT), Trails A and B, Brief Visuospatial Memory Test (BVMT), Stroop Test, Wechsler Test of Adult Reading (WTAR), Brief Test of Attention, (BTA), Wisconsin Card Sorting Test (WCST) and COWAT (Controlled Oral Word Association Test). The WTAR will be used as an estimate of IQ and the neurocognitive test T-scores of interest will be compared against the subject's IQ T-score. The standard deviation (SD) of each T-score is 10. Each of the subject's neurocognitive tests is considered aberrant if it is more than 2 SD below the subject's IQ T-score. A subject is considered cognitively impaired if at least 2 (based on the .05 rule; 5 out of every 100 test scores will be outside of expected range by chance alone) out of the T-scores are aberrant.
Time Frame: 3 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Moderate/Severe Post-Concussive Symptoms
Description: Moderate/severe post-concussive symptoms will be defined as the presence of any one or more of the following: headaches, dizziness, general malaise, excessive fatigue, or noise intolerance, irritability, emotional lability, depression, or anxiety, subjective complaints of concentration or memory difficulty, insomnia, reduced tolerance to alcohol, preoccupation with these symptoms and fear of permanent brain damage. These will be self-reported by the patient.
Time Frame: 3 months
Reporting Status: Not Posted

9. Post Hoc Outcome: Glial Fibrillary Acidic Protein (GFAP)
Time Frame: 3 months
Population: Missing blood samples due to loss of follow-up.
Measure: Mean (Inter-Quartile Range); unit: picograms per ml
Arm/Group | Omega-3 Polyunsaturated Fatty Acid Treatment Arm | Placebo Arm
Number analyzed (Participants) | 19 | 19
picograms per ml
  Baseline | 77.9 [56.8 to 158.0] | 53.7 [40.4 to 123.0]
  1 month: number analyzed (Participants) | 14 | 10
  1 month | 51.0 [41.3 to 91.0] | 87.7 [59.6 to 118.8]
  3 month: number analyzed (Participants) | 12 | 8
  3 month | 61.2 [31.2 to 99.7] | 68.4 [45.7 to 129.0]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Omega-3 Polyunsaturated Fatty Acid Treatment Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 3/22 | 0/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 Polyunsaturated Fatty Acid Treatment Arm (N=22) | Placebo Arm (N=22)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT03345550/Prot_SAP_000.pdf